CLINICAL TRIAL: NCT03937700
Title: Robot Based Gait Training Therapy for Pediatric Population With Cerebral Palsy Using the CPWalker
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Arun Jayaraman, PT, PhD, Research Scientist, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00206310
Record Dates: First submitted 2019-05-01; First posted 2019-05-06 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPWalker Robotic-Assisted Gait Training (Experimental): Each subject will participate in 16-24 gait training sessions in the CPWalker over the course of 8 weeks with each session lasting up to 2 hours
  Interventions: Device: CPWalker Robotic Exoskeleton

INTERVENTIONS:
Device: CPWalker Robotic Exoskeleton — The CPWalker rehabilitation platform is a robotic device composed by an exoskeleton linked to a walker that provides support and balance to a child during overground training. The device is able to implement user's partial body weight support (PBWS) and allows the adaptation of exercises to the patient's capabilities by means of individual controllers for each joint, which increases the modularity of the system. Each joint of the CPWalker can operate in a range of modes with varied levels of robotic assistance or resistance

SUMMARY:
This trial is being conducted to determine if the CPWalker can be used as a gait training intervention for pediatric patients with gait impairments due to cerebral palsy

DETAILED DESCRIPTION:
Objectives:

1. To determine the use of the CPWalker rehabilitation platform, a robotic device composed by an exoskeleton linked to a walker that provides support and balance, as a gait training intervention in the pediatric cerebral palsy population.
2. To create and define detailed guidelines consisting of robotic based treatment methods for gait rehabilitation.

Hypothesis:

1. CPWalker can be used as a gait training intervention for pediatric patients with gait impairments due to cerebral palsy
2. Performing lower limb training in conjunction with active head and trunk control therapies will improve functional gait levels
3. Following 16-24 CPWalker training sessions, persons with cerebral palsy will show improvements in functional mobility when comparing pre-training measurements to post-training measurements

Procedures:

Participants will engage in an 8-week training program, consisting of 2-3 sessions per week based on the level of gait impairment. Percentage range of motion (ROM), partial body weight support (PWBS), and gait velocity are the principal parameters under variation during training.

Additionally, screening, baseline and post-training testing sessions will be conducted

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Cerebral Palsy with spastic diplegia
* Gross Motor Function Classification System score of 2-4
* Age 11-21 at time of enrollment
* Maximum weight of 75kg
* Height range of approximately 110cm to 170cm
* Ability to understand and follow verbal cues
* Lower limb measurements meet specifications of CPWalker
* Cognition sufficient to communicate pain or discomfort and follow one step direction from the investigator

Exclusion Criteria:

* Any orthopedic surgeries less than 3 months prior to study enrollment or ongoing botox injections
* Severe musculoskeletal deformities affecting safe and comfortable fit into the exoskeleton as determined by the investigator. Patients may be able to wear their AFOs in the CPWalker if it allows for safe fit.
* Unhealed wounds/lesions
* Critical motor control alterations such as dystonia, choreoathetosis, or ataxia
* Aggressive or self-harming behavior
* Severe cognitive impairments that prevent a subject from being able to understand the exercises an/or interact with the study staff

Ages: 11 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
10-Meter Walk Test | Change from baseline gait speed at 8 weeks
  This test will examine the patient's gait speed. Patients will be directed to walk at their preferred and maximum but safe speed. Patients will be positioned 1 meter before the start line and instructed to walk the entire 10-meter distance and past the end line approximately 1 meter. The distance before and after the course are meant to minimize the effect of acceleration and deceleration. Time will be recorded using a stopwatch and recorded to the one hundredth of a second.

SECONDARY OUTCOMES:
6-Minute Walk Test | Change from baseline distance ambulated at 8 weeks
  This test measures the distance a subject can walk indoors on a flat, hard surface in a period of 6 minutes, using assistive devices, as necessary. The test is a reliable and valid evaluation of functional exercise capacity and is used as a sub-maximal test of aerobic capacity and endurance. The test is patient self-paced and assesses the level of functional capacity. Patients are allowed to stop and rest during the test, however, the timer does not stop. If the patient is unable to complete the time, the time stopped is noted and reason for stopping prematurely is recorded. This test will be administered while wearing a mask to measure oxygen consumption.
GAITRite Data Collection | Change from baseline gait quality at 8 weeks
  The GAITRite system automates measuring temporal and spatial gait parameters via an electronic walkway connected to a computer. The GAITRite electronic walkway contains sensor pads encapsulated in a carpet to collect gait information. The system can be laid over any flat surface. The GAITRite electronic walkway for the study shall be a minimum of 14 feet long. The GAITRite data capture was chosen as measurement of the patient's overall gait quality. Patients will be asked to walk at a self-selected speed across the GAITRite electronic walkway with at least a two meter "flying start" to compensate for initial acceleration.
Pediatric Balance Scale | Change from baseline balance score at 8 weeks
  This test is a 14-item objective measure designed to assess static balance in pediatric populations. The functional activities that are assessed include sitting and standing balance during transfers, altered base of support, reaching, turning, eyes open and closed. Each item is scored from 0 to 4 points. The maximum score is 56 points.
Selective Control Assessment of Lower Extremity (SCALE) | Change from baseline selective voluntary motor control at 8 weeks
  This clinical tool quantifies selective voluntary motor control of the lower extremities in patients with cerebral palsy.
Gross Motor Function Measure (GMFM-88) dimensions D (standing) and E (walking) | Change from baseline gross motor function at 8 weeks
  This test measures the change in gross motor function with intervention in children with cerebral palsy
Child and Adolescent Scale of Participation | Change in children's baseline participation in activities at 8 weeks
  This questionnaire measures the extent to which children participate in home, school, and community activities as reported by family caregivers.
Gillette Functional Assessment Questionnaire (FAQ) | Change in baseline report of ambulatory function at 8 weeks
  This is a proxy-report measure that includes a ten-level classification of ambulatory function and 22 functional locomotor activities

CONTACTS AND LOCATIONS:
Overall Officials: Arun Jayaraman, PT, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States